CLINICAL TRIAL: NCT05857501
Title: Preoperative Prediction of Flexible Ureteroscopy Outcome in the Treatment of Renal Calculi
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, islam mohamed abou bakr mansour, Teaching Assistant, Menoufia University
Other Study IDs: FURS outcome prediciton
Record Dates: First submitted 2023-04-10; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Flexible Ureteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: abdominopelvic computerized tomography (CT) without contrast — scan combines a series of X-ray images taken from different angles around your body and uses computer processing to create cross-sectional images (slices) of the bones, blood vessels and soft tissues inside your body. CT scan images provide more-detailed information than plain X-rays do.
  Other Names: digital KUB (plain x-ray on urology system )

SUMMARY:
To predict the outcome of flexible ureteroscopy in the management of renal stones based on preoperative scoring module using five preoperative parameters that have effect on stone free status postoperatively.

DETAILED DESCRIPTION:
Although flexible ureteroscopy has been in use for decades, neither the European Association of Urology (EAU) nor the American Urological association (AUA), in their clinical guidelines, recommends flexible ureteroscopy (FURS) as a first-line procedural treatment for renal stones . Several reports showed that FURS is a suitable alternative to shockwave lithotripsy (SWL) and percutaneous nephrolithotripsy (PCNL) for the treatment of renal stones, with potentially higher stone-free rates than SWL and lower morbidity than PCNL.

Safe and effective removal by FURS of multiple and large intrarenal stones, including lower pole calculi, has been documented suggesting that FURS is effective for complex intrarenal stone removal . With the multitude of available procedures, selection of the optimal one for management of renal stone is becoming more challenging.

Established models for predicting the outcomes of SWL and PCNL exist . However, a predictive model for predicting the outcome of URS is still in development , particularly for FURS treatment of renal stones. Four scores have been developed for FURS. Two of these have been compared and validated in different cohorts: the Resolu Unsal Stone Score (RUSS) and modified Seoul National University Renal Stone Complexity (S-ReSC) score , the other two scores, the S.T.O.N.E score described by Molina et al. and Ito's nomogram.

Many studies have demonstrated that stone volume is the most significant factor predictive of stone-free status (SF) after FURS. The investigators speculate that stone volume combined with other variables might improve prediction of SF after FURS. The aim of the present study is to evaluate various preoperative parameters as predictors of FURS outcome based on the Ito's nomogram

ELIGIBILITY:
Inclusion Criteria:

1. Renal stones (≤ 2 cm)
2. Radiolucent stone resistant to SWL and oral chemical dissolution treatment (≤2cm)

Exclusion Criteria:

1. Large stones (> 2 cm).
2. Staghorn stone (stone involving the renal pelvis and more than two calyces).
3. Patient preference of other treatment modality

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with renal stones that are < 2 cm in maximal diameter will be recruited to the study. Patients will be counseled for flexible ureteroscopy, and the procedure will be explained to them with discussion about its pros and cons. Patients agreeable to enrollment will sign an informed written consent after fulfillment of ethical approval forms.Stone free rate will be assessed at one week, one month, and three months post-operatively using Plain X-ray for radio-opaque stones and NCCT for radiolucent stones.
  Stone free rate will be determined by no stone fragment > 4mm. Number of ancillary procedures required to reach SF will be reported
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
stone free rate after flexible ureteroscopy | baseline
  the investigators predict the outcome of flexible ureteroscopy in the management of renal stones based on preoperative scoring module using five preoperative parameters that have effect on stone free rate postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelgaber Selim, ASS-PROF, Principal Investigator — menofia universtiy

REFERENCES:
- [Background] Preminger GM, Tiselius HG, Assimos DG, Alken P, Buck C, Gallucci M, Knoll T, Lingeman JE, Nakada SY, Pearle MS, Sarica K, Turk C, Wolf JS Jr; EAU/AUA Nephrolithiasis Guideline Panel. 2007 guideline for the management of ureteral calculi. J Urol. 2007 Dec;178(6):2418-34. doi: 10.1016/j.juro.2007.09.107. No abstract available. PMID 17993340
- [Background] Tiselius HG, Ackermann D, Alken P, Buck C, Conort P, Gallucci M; Working Party on Lithiasis, European Association of Urology. Guidelines on urolithiasis. Eur Urol. 2001 Oct;40(4):362-71. doi: 10.1159/000049803. PMID 11713390
- [Background] El-Nahas AR, Ibrahim HM, Youssef RF, Sheir KZ. Flexible ureterorenoscopy versus extracorporeal shock wave lithotripsy for treatment of lower pole stones of 10-20 mm. BJU Int. 2012 Sep;110(6):898-902. doi: 10.1111/j.1464-410X.2012.10961.x. Epub 2012 Feb 28. PMID 22372915
- [Background] Cohen J, Cohen S, Grasso M. Ureteropyeloscopic treatment of large, complex intrarenal and proximal ureteral calculi. BJU Int. 2013 Mar;111(3 Pt B):E127-31. doi: 10.1111/j.1464-410X.2012.11352.x. Epub 2012 Jul 3. PMID 22757752
- [Background] Pearle MS, Lingeman JE, Leveillee R, Kuo R, Preminger GM, Nadler RB, Macaluso J, Monga M, Kumar U, Dushinski J, Albala DM, Wolf JS Jr, Assimos D, Fabrizio M, Munch LC, Nakada SY, Auge B, Honey J, Ogan K, Pattaras J, McDougall EM, Averch TD, Turk T, Pietrow P, Watkins S. Prospective randomized trial comparing shock wave lithotripsy and ureteroscopy for lower pole caliceal calculi 1 cm or less. J Urol. 2008 May;179(5 Suppl):S69-73. doi: 10.1016/j.juro.2008.03.140. PMID 18405758
- [Background] Akman T, Binbay M, Ozgor F, Ugurlu M, Tekinarslan E, Kezer C, Aslan R, Muslumanoglu AY. Comparison of percutaneous nephrolithotomy and retrograde flexible nephrolithotripsy for the management of 2-4 cm stones: a matched-pair analysis. BJU Int. 2012 May;109(9):1384-9. doi: 10.1111/j.1464-410X.2011.10691.x. Epub 2011 Oct 28. PMID 22093679
- [Background] Breda A, Ogunyemi O, Leppert JT, Schulam PG. Flexible ureteroscopy and laser lithotripsy for multiple unilateral intrarenal stones. Eur Urol. 2009 May;55(5):1190-6. doi: 10.1016/j.eururo.2008.06.019. Epub 2008 Jun 13. PMID 18571315
- [Background] Breda A, Ogunyemi O, Leppert JT, Lam JS, Schulam PG. Flexible ureteroscopy and laser lithotripsy for single intrarenal stones 2 cm or greater--is this the new frontier? J Urol. 2008 Mar;179(3):981-4. doi: 10.1016/j.juro.2007.10.083. Epub 2008 Jan 22. PMID 18207179
- [Background] Takazawa R, Kitayama S, Tsujii T. Successful outcome of flexible ureteroscopy with holmium laser lithotripsy for renal stones 2 cm or greater. Int J Urol. 2012 Mar;19(3):264-7. doi: 10.1111/j.1442-2042.2011.02931.x. Epub 2011 Dec 6. PMID 22145599
- [Background] Wiesenthal JD, Ghiculete D, Ray AA, Honey RJ, Pace KT. A clinical nomogram to predict the successful shock wave lithotripsy of renal and ureteral calculi. J Urol. 2011 Aug;186(2):556-62. doi: 10.1016/j.juro.2011.03.109. PMID 21684557
- [Background] Kanao K, Nakashima J, Nakagawa K, Asakura H, Miyajima A, Oya M, Ohigashi T, Murai M. Preoperative nomograms for predicting stone-free rate after extracorporeal shock wave lithotripsy. J Urol. 2006 Oct;176(4 Pt 1):1453-6; discussion 1456-7. doi: 10.1016/j.juro.2006.06.089. PMID 16952658
- [Background] Smith A, Averch TD, Shahrour K, Opondo D, Daels FP, Labate G, Turna B, de la Rosette JJ; CROES PCNL Study Group. A nephrolithometric nomogram to predict treatment success of percutaneous nephrolithotomy. J Urol. 2013 Jul;190(1):149-56. doi: 10.1016/j.juro.2013.01.047. Epub 2013 Jan 23. PMID 23353048
- [Background] Imamura Y, Kawamura K, Sazuka T, Sakamoto S, Imamoto T, Nihei N, Suzuki H, Okano T, Nozumi K, Ichikawa T. Development of a nomogram for predicting the stone-free rate after transurethral ureterolithotripsy using semi-rigid ureteroscope. Int J Urol. 2013 Jun;20(6):616-21. doi: 10.1111/j.1442-2042.2012.03229.x. Epub 2012 Nov 19. PMID 23163835
- [Background] Resorlu B, Unsal A, Gulec H, Oztuna D. A new scoring system for predicting stone-free rate after retrograde intrarenal surgery: the "resorlu-unsal stone score". Urology. 2012 Sep;80(3):512-8. doi: 10.1016/j.urology.2012.02.072. Epub 2012 Jul 26. PMID 22840867
- [Background] Jung JW, Lee BK, Park YH, Lee S, Jeong SJ, Lee SE, Jeong CW. Modified Seoul National University Renal Stone Complexity score for retrograde intrarenal surgery. Urolithiasis. 2014 Aug;42(4):335-40. doi: 10.1007/s00240-014-0650-7. Epub 2014 Mar 13. PMID 24623504
- [Background] Molina WR, Kim FJ, Spendlove J, Pompeo AS, Sillau S, Sehrt DE. The S.T.O.N.E. Score: a new assessment tool to predict stone free rates in ureteroscopy from pre-operative radiological features. Int Braz J Urol. 2014 Jan-Feb;40(1):23-9. doi: 10.1590/S1677-5538.IBJU.2014.01.04. PMID 24642147
- [Background] Ito H, Sakamaki K, Kawahara T, Terao H, Yasuda K, Kuroda S, Yao M, Kubota Y, Matsuzaki J. Development and internal validation of a nomogram for predicting stone-free status after flexible ureteroscopy for renal stones. BJU Int. 2015 Mar;115(3):446-51. doi: 10.1111/bju.12775. Epub 2014 Aug 13. PMID 24731157
- [Background] Ito H, Kawahara T, Terao H, Ogawa T, Yao M, Kubota Y, Matsuzaki J. Utility and limitation of cumulative stone diameter in predicting urinary stone burden at flexible ureteroscopy with holmium laser lithotripsy: a single-center experience. PLoS One. 2013 Jun 4;8(6):e65060. doi: 10.1371/journal.pone.0065060. Print 2013. PMID 23750229
- [Background] Ito H, Kawahara T, Terao H, Ogawa T, Yao M, Kubota Y, Matsuzaki J. The most reliable preoperative assessment of renal stone burden as a predictor of stone-free status after flexible ureteroscopy with holmium laser lithotripsy: a single-center experience. Urology. 2012 Sep;80(3):524-8. doi: 10.1016/j.urology.2012.04.001. Epub 2012 Jun 1. PMID 22658621